CLINICAL TRIAL: NCT03435978
Title: Effect of Three-month Diet and Physical Activity on Adipokines and Inflammatory Status in Children With Metabolic Syndrome
Brief Title: Effect of Diet and Physical Activity on Adipokines
Status: Completed | Type: Observational
Sponsor: Louis Turcanu Emergency Hospital for Children (Other)
Collaborators: University of Medicine and Pharmacy "Victor Babes" Timisoara (Other)
Responsible Party: Principal Investigator, Ramona Stroescu, MD,PhD,Clinical Researcher, Louis Turcanu Emergency Hospital for Children
Other Study IDs: 13200
Record Dates: First submitted 2018-01-31; First posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Obesity, Metabolically Benign
Keywords: diet; metabolic syndrome; obese children
MeSH Terms: conditions — Obesity, Metabolically Benign; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MetS+: Obese group with metabolic syndrome/Data processing from Patient Medical Files
  Interventions: Behavioral: MetS+
- MetS-: Obese group without metabolic syndrome/Data processing from Patient Medical Files
  Interventions: Other: MetS-

INTERVENTIONS:
Behavioral: MetS+
  Groups: MetS+
Other: MetS- — Data processing from Patient Medical Files
  Groups: MetS-

SUMMARY:
The prevalence of metabolic syndrome (MetS) in young population continues to rise. Obesity is a chronic inflammatory disorder in which leptin, adiponectin and C reactive protein (CRP) play an important role. This study aimed to determine whether these adipokines are significant markers in defining MetS in pediatric population and to assess the effect of hypocaloric diet and physical activity on serum concentrations of adiponectine, leptin, and high sensitivity CRP (hs-CRP).

DETAILED DESCRIPTION:
The idea that adipose tissue is just a form of energy storage has changed dramatically in recent years. Currently, adipose tissue is considered to be a true endocrine gland that fulfills multiple roles in regulating different biological functions. Communication between adipose tissue and the rest of the systems is accomplished through bioactive mediators (adipokines) Adipokines control energy homeostasis and are involved in metabolic, endocrine and immunological processes.The prevalence of metabolic syndrome (MetS) in young population continues to rise. Obesity is a chronic inflammatory disorder in which leptin, adiponectin and C reactive protein (CRP) play an important role. This study aimed to determine whether these adipokines are significant markers in defining MetS in pediatric population and to assess the effect of hypocaloric diet and physical activity on serum concentrations of adiponectine, leptin, and high sensitivity CRP (hs-CRP).

The investigators tested the hypothesis that long-term lifestyle changes and moderate weight loss would reduce the plasma concentrations of adipokines involved in inflammation, angiogenesis, and chemotaxis and would increase adiponectin concentrations.

Material and methods:

A prospective study was conducted over a period of 1 year, between January 2016 and December 2016, on 66 cases of obesity in children diagnosed at the Louis Ţurcanu Emergency Hospital for Children Timisoara. The patients diagnosed with MetS were put on diet and physical exercise for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* obese children (BMI> 95th percentile)

Exclusion Criteria:

* obesity caused by endocrine disease, syndromic obesity, systemic disease or acute illness.

Ages: 5 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: All children admitted to the Endocrinology, Diabetology and Cardiology Department who met the Inclusion Criteria
Sampling Method: Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2018-01-03 (Actual)

PRIMARY OUTCOMES:
Defining obesity in the pediatric population | Weight and height were measured on day 1 of admission. Obesity was defined as a BMI > the 95th percentile.
  Measuring weight in kilograms and height in meters in order to calculate BMI and represent it on the percentile graph.
Leptin changes in the obese children with metabolic syndrome | Leptin levels were measured on day 1 of admission and after three months. Normal range was considered < 24ng/ml.
  Evaluating leptin in the obese group with metabolic syndrome after three months of diet and physical activity.
Adiponectin changes in the obese children with metabolic syndrome | Adiponectin levels were measured on day 1 of admittance and after three months in children aged between 4 and 18 years. Levels 4-26 mcg/ml were defined as normal values.
  Evaluating adiponectin in the obese group with metabolic syndrome after three months of diet and physical activity.
hsCRP changes in the obese children with metabolic syndrome | hsCRP levels were measured on day 1 of admittance and after three months in children aged between 4 and 18 years. Normal levels were considered between 0.1-2.8 mg/l.
  Evaluating hsCRP in the obese group with metabolic syndrome after three months of diet and physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Mihai Gafencu, Md,PhD, Principal Investigator — Louis Turcanu Emergency Hospital for Children

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beyazit F, Unsal MA. Obesity and insulin resistance are significant predictors of serum leptin levels. J Turk Ger Gynecol Assoc. 2017 Sep 1;18(3):158-159. doi: 10.4274/jtgga.2017.0027. No abstract available. PMID 28890432
- [Background] Bagherniya M, Khayyatzadeh SS, Heidari Bakavoli AR, Ferns GA, Ebrahimi M, Safarian M, Nematy M, Ghayour-Mobarhan M. Serum high-sensitive C-reactive protein is associated with dietary intakes in diabetic patients with and without hypertension: a cross-sectional study. Ann Clin Biochem. 2018 Jul;55(4):422-429. doi: 10.1177/0004563217733286. Epub 2017 Nov 23. PMID 28882065